CLINICAL TRIAL: NCT02251652
Title: An Investigator-Initiated Study to Assess the Safety and Efficacy of Ingenol Mebutate 0.05% Gel When Used After Cryotherapy in the Treatment of Hypertrophic Actinic Keratoses (AK) on Dorsal Hands
Brief Title: Safety and Efficacy of Ingenol Mebutate 0.05% Gel When Used After Cryotherapy in the Hypertrophic Actinic Keratoses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Gary Goldenberg, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 13-0142
Record Dates: First submitted 2014-09-17; First posted 2014-09-29 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Actinic Keratoses
Keywords: Actinic
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Therapy (Active Comparator): Cryotherapy followed by Ingenol Mebutate Gel
  Interventions: Drug: Ingenol Mebutate; Procedure: Cryotherapy
- Cryotherapy Alone (Active Comparator): Cryotherapy only
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Drug: Ingenol Mebutate — Ingenol mebutate 0.05% gel
  Other Names: PEP005 Gel
  Arms: Combination Therapy
Procedure: Cryotherapy — 1-2 sprays, 5 seconds each, with a 5 second interval

SUMMARY:
Sequential therapy with cryosurgery and ingenol mebutate may optimize the treatment of hypertrophic AKs and also treat non-hypertrophic AKs in this anatomic location. Furthermore, use of ingenol mebutate will also be evaluated for potential treatment of subclinical lesions.

DETAILED DESCRIPTION:
The investigators plan to treat 30 subjects. Each qualifying subject will have at least 3 hypertrophic AKs, defined as more than 3mm in thickness, on each dorsal hand. Cryotherapy will be standardized in all patients and for all treated lesions: 1-2 sprays, 5 seconds each, with a 5 second interval. All subjects will be treated with the same cryo-spray. Following cryotherapy, subjects will be randomized to treat either their right or left dorsal hand with ingenol mebutate gel. The decision to treat the right vs. the left hand will be chosen by chance, like flipping a coin. Neither the subject nor the study doctor will choose what arm receives the ingenol mebutate gel. The study doctor will not know which arm is treated with ingenol mebutate, so the subject should not reveal that information to him or her at any time during the study. Subjects will treat the randomized dorsal hand with ingenol mebutate 0.05% gel starting on the same day as the cryotherapy (Day 0). Subjects will utilize the once daily for two days regimen. Subjects will be followed on day 4 after their initial visit, day 8, day 15, day 29, and day 57, with a two day window period.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old.
* Subjects must be in good general health as confirmed by the medical history.
* Subjects must be able to read, sign, and understand the informed consent
* Prior to cryosurgery, subjects have at least 3 hypertrophic actinic keratoses on each dorsal hand.
* Subject must be willing to forego any other treatments on the dorsum of the hands, including tanning bed use and excessive sun exposure while in the study.
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and to comply with all study requirements including concomitant medication and other treatment restrictions.
* If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study.

Exclusion Criteria:

* Subjects with a history of melanoma anywhere on the body.
* Subjects with an unstable medical condition as deemed by the clinical investigator.
* Subjects with non-melanoma skin cancer on the dorsum of the hands.
* Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of AKs.
* Subjects who have previously been treated with ingenol mebutate: on the dorsum of the hands in the past 6 months; or outside of the study area within the past 30 days.
* Women who are pregnant, lactating, or planning to become pregnant during the study period.
* Subjects who have experienced a clinically important medical event within 90 days of the visit (e.g., stroke, myocardial infarction, etc).
* Subjects who have active chemical dependency or alcoholism as assessed by the investigator.
* Subjects who have known allergies to any excipient in the study gel.
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device on the study area within 30 days prior to study treatment initiation.
* Subjects who have received any of the following within 90 days prior to study treatment initiation:

  * interferon or interferon inducers
  * cytotoxic drugs
  * immunomodulators or immunosuppressive therapies (inhaled/ intranasal steroids are permitted)
  * oral or parenteral corticosteroids
  * topical corticosteroids if greater than 2 gm/day
  * any dermatologic procedures or surgeries on the study area (including any AK treatments)
* Subjects who have used any topical prescription medications on the study area within 30 days prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Goldenberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Hashim PW, Nia JK, Singer S, Goldenberg G. An Investigator-initiated Study to Assess the Safety and Efficacy of Ingenol Mebutate 0.05% Gel When Used After Cryosurgery in the Treatment of Hypertrophic Actinic Keratosis on Dorsal Hands. J Clin Aesthet Dermatol. 2016 Jul;9(7):16-22. Epub 2016 Jul 1. PMID 27672408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Faculty Practice and resident clinics at Mount Sinai. Seventeen subjects were enrolled in the study; one subject withdrew consent prior to treatment.
Groups:
- Actinic Keratosis: Each subject is its own control - left dorsal hand compared to right dorsal hand
Period: Overall Study
Arm/Group | Actinic Keratosis
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Actinic Keratosis
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.06 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Safety of Combination Therapy vs Cryotherapy Alone
Description: To evaluate the safety of cryotherapy plus ingenol mebutate on dorsal hands and compare it to the safety of cryotherapy alone looking at Adverse Events.
Time Frame: Day 57
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy | Cryotherapy Alone
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

2. Secondary Outcome: Change in Number of All Actinic Keratoses
Description: To evaluate and compare the mean reduction in number of all AKs (hypertrophic and non-hypertrophic) on the dorsal hands of the combination cryotherapy- ingenol mebutate treated side vs. the cryotherapy alone side on Day 57 as compared to baseline
Time Frame: Baseline and Day 57
Population: Comparisons of proportion of responders between treated and control hands
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: Actinic Keratoses lesions
Arm/Group | Combination Therapy | Cryotherapy Alone
Number analyzed (Participants) | 16 | 16
Number analyzed (Actinic Keratoses lesions) | 73 | 87
percent change | -4.6 (2.66) | -2.5 (1.37)

3. Secondary Outcome: Change in Actinic Keratoses by Anatomic Site
Description: To evaluate the number of AKs (both hypertrophic and non-hypertrophic) before therapy by anatomic site (dorsal hand) at Day 57 as compared to baseline
Time Frame: Baseline and Day 57
Population: Comparisons of proportion of responders between treated and control hands
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: Actinic Keratoses lesions
Arm/Group | Combination Therapy | Cryotherapy Alone
Number analyzed (Participants) | 16 | 16
Number analyzed (Actinic Keratoses lesions) | 73 | 87
percent change
  Hypertrophic | -86.34 (16.642) | -51.89 (19.091)
  Non-hypertrophic | -4.1 (3.38) | 0.0 (0.0)

ADVERSE EVENTS:
Arm/Group | Combination Therapy | Cryotherapy Alone
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
Study limitations include small sample size and the fact that LSRs may unblind the investigator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes